CLINICAL TRIAL: NCT00083434
Title: Treatment of Anemic Patients With Cancer Who Are Not Receiving Chemotherapy or Radiotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped because of an inadequate rate of enrollment.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Purpose: Treatment
Other Study IDs: CR010549; EPO-CAN-303
Record Dates: First submitted 2004-05-24; First posted 2004-05-26 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Anemia; Cancer
Keywords: Anemia; Cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to examine the effectiveness of epoetin alfa in treating anemia in patients who have cancer or who no longer have any signs of the cancer, but remain anemic as a result of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body weight >/= 99lbs
* ECOG 0-2
* Anemia results from cancer, chemotherapy, radiotherapy or an association with hormonal therapy or immunotherapy
* Screening hemoglobin level of </= 11.0 g/dL for men or </= 10.0 for women

Exclusion Criteria:

* History of or concurrent second malignancy
* Evidence of primary or metastatic malignancy involving the Central Nervous System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Advanced Urology Medical Center, Anaheim, California
  - Shapiro, Stafford & Yee, Arcadia, California
  - California Cancer Center, Fresno, California
  - Tukoi Research, North Miami, Florida
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Madigan Army Medical Center Urology Services, Tacoma, Washington

REFERENCES:
- See also: FDA Approved Product labeling, refer to the following link:http://www.accessdata.fda.gov/scripts/cder/drugsatfda/ — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/
- See also: Additional information is provided at the following link:http://dailymed.nlm.nih.gov/dailymed/about.cfm — http://dailymed.nlm.nih.gov/dailymed/about.cfm